CLINICAL TRIAL: NCT00581633
Title: Acute Renal Salt Handling in Orthostatic Intolerance
Brief Title: Acute Salt Handling in Orthostatic Intolerance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Satish R. Raj, Assistant Professor of Medicine & Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 061230; UL1RR024975 (NIH); K23RR020783 (NIH); P01HL056693 (NIH)
Record Dates: First submitted 2007-12-22; First posted 2007-12-27 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Postural Tachycardia Syndrome; Orthostatic Tachycardia; Orthostatic Intolerance
Keywords: saline; sodium; kidney; tachycardia
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance; Tachycardia | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): saline infusion for sodium loading
  Interventions: Other: normal saline (0.9%)

INTERVENTIONS:
Other: normal saline (0.9%) — liter normal saline over 30 minutes x 1 dose

SUMMARY:
The investigators will test the hypothesis that patients with chronic orthostatic intolerance or postural orthostatic tachycardia syndrome (OI or POTS) will be unable to conserve urinary sodium as compared to healthy control subjects.

DETAILED DESCRIPTION:
Patients with chronic OI appear to be hypovolemic with abnormalities in hormones that regulate salt & water handling. Increases in dietary salt have salutary effects on orthostatic tolerance in a physiological laboratory. The infusion of intravenous saline acutely decreased heart rate in this patient population. Preliminary data from Vanderbilt suggests abnormal salt handling in patients with chronic OI in a few patients. These data need to be confirmed and a better understanding of sodium handling in response to acute salt loads is required in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with orthostatic intolerance by Vanderbilt Autonomic Dysfunction Center (or healthy control subject)

Exclusion Criteria:

* Overt or acute cause for orthostatic tachycardia
* Hypertension (BP>145/95 or need for anti-hypertensive medications)
* QRS duration > 120 msec on EKG
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-02; Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Urinary Na excretion | 24h and then hourly post saline load

SECONDARY OUTCOMES:
Catecholamine levels | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt Autonomic Dysfunction Center — https://www.vumc.org/autonomic-dysfunction-center/vanderbilt-autonomic-dysfunction